CLINICAL TRIAL: NCT06783543
Title: Efficacy of Home-based Treatment for Breast Cancer-related Lymphedema
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: yan2024-1125
Record Dates: First submitted 2025-01-05; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Lymphedema Arm
Keywords: lymphedema; breast cancer; Manual therapy; home-based therapy
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: According to the computer random number method, the enrolled patients were divided into home treatment group and outpatient treatment group, 20 cases each.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- home-based group (Experimental): In this group of patients, the therapist conducted standardized comprehensive detumescence treatment at the first treatment which including four steps of skin care, manual lymphatic drainage, low-elastic bandage dressing and functional exercise. After the treatment, videos of manual lymphatic drainage and pressure dressing of family members were provided. Patients or family members were required to perform this treatment at home every day. Video recordings were necessary during treatment at home which were required be sent to the therapist, making sure the session is done every day. They returned to the edema clinic one month later for another evaluation. If patients encounter problems that cannot be solved during home treatment, they should consult online on wechat, or return to the edema clinic in time.
  Interventions: Other: Comprehensive detumescence treatment with education video
- outpatient group (Active Comparator): Patients were required to go to the lymphedema clinic for comprehensive detumescence treatment, including skin care, manual lymphatic drainage, low-elastic bandaging and functional exercise, 3 to 5 times a week for 1 hour each time. They were re-evaluated after one month of treatment.
  Interventions: Other: Comprehensive detumescence treatment

INTERVENTIONS:
Other: Comprehensive detumescence treatment with education video — Comprehensive detumescence treatment, including skin care, manual lymphatic drainage, low elastic bandaging and functional exercise four steps
  Other Names: Education video of manual lymphatic drainage and pressure bandaging
  Arms: home-based group
Other: Comprehensive detumescence treatment — Three to five times a week, one hour each time
  Arms: outpatient group

SUMMARY:
The goal of this clinical trials is to explore the effectiveness of home-based iymphedema treatment and the differences between the home-based and outpatient treatment. The main question is to verify that home-based treatment is as effective as outpatient treatment. We set two groups in this study, comparing the volume of affected upper limb to see if home-based iymphedema treatment is valuable method.

DETAILED DESCRIPTION:
Secondary outcome measures:

1. Core Quality of Life Questionnaire (EORTC QLQ-C30), It included five functional measures (somatic function, role function, cognitive function, emotional function, social function), three symptom measures (fatigue, pain, nausea and vomiting), six individual measures (dysphagia, loss of appetite, sleep disturbance, constipation, diarrhea, financial hardship), and one patient self-assessment item (total health status).
2. Breast Cancer and Lymphedema Symptom Experience Index (BCLE-SEI).

ELIGIBILITY:
Inclusion Criteria:

1. Lymphedema appeared in the upper limb after breast cancer-related treatment, and compared with the healthy side, the edema dimension was more than 2cm.
2. Age 18-75 years old;
3. Edema stage Ⅰ to Ⅱ;

Exclusion Criteria:

1. People with severe cognitive impairment;
2. Bilateral lymphedema;
3. Patients undergoing radiotherapy；
4. Patients with uncontrolled tumors;
5. Congestive heart failure and other comprehensive detumescence treatment contraindicated patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-11-13 (Estimated); Study Completion 2025-12-13 (Estimated)

PRIMARY OUTCOMES:
the volum of affected arm | at the first day and after one month
  A soft ruler was used to measure the patient's wrist stripes and 10cm, 20cm, 30cm and 40cm above the wrist stripes, respectively, to obtain the circumference value. The five measurement points can divide the limb into four truncated cones, and then the formula can be used to calculate the volume of each limb segment, in which C1 and C2 are the arm circumference of the upper and lower two points of the measurement segment. h is the length of the measuring section, that is, 10 cm, and the whole limb volume is the sum of the volumes of each section.

SECONDARY OUTCOMES:
Quality of life Core questionnaire scale -- EORTC QLQ-C30 | at the first day and after one month
  It included five functional measures (somatic function, role function, cognitive function, emotional function, social function), three symptom measures (fatigue, pain, nausea and vomiting), six individual measures (dysphagia, loss of appetite, sleep disturbance, constipation, diarrhea, financial hardship), and one patient self-assessment item (total health status).
Breast Cancer and Lymphedema Symptom Experience Index， BCLE-SEI | at the first day and after one month

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
The primary outcome mesurement will be shared.